CLINICAL TRIAL: NCT02375984
Title: A Phase II Study Using Tumor-Reactive Autologous Tumor Infiltrating Lymphocytes (TIL) Plus IL-2 Followed by Lymphocyte Depleting Chemotherapy Regimen in Metastatic Melanomas
Brief Title: A Study Using Tumor-Reactive Autologous Tumor Infiltrating Lymphocytes (TIL) in Metastatic Melanomas
Acronym: TIL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI changed institutions
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIL-TREATMENT-0614
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tumor Infiltrating Lymphocytes (TIL) (Experimental): Patients will have a melanoma metastasis resected and cultured in IL-2 in vitro either as part of this treatment protocol or the JWCI procurement protocol. TIL from these cultures will be assessed for tumor-reactivity and those with such activity will be further expanded and adoptively transferred. Patients will receive a non-myeloablative lymphocyte-depleting preparative regimen consisting of cyclophosphamide (60 mg/kg/day X 2 days IV) and fludarabine (25 mg/m2/day IV X 5 days). Following this regimen, patients will receive an intravenous adoptive transfer of at least 109 tumor-reactive lymphocytes (TIL) followed by high-dose intravenous IL-2 (600-720,000 IU/kg/dose every 8 hours for up to 12 doses).
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — Patients will receive an IV adoptive transfer of at least 10^9 tumor-reactive lymphocytes. An IV catheter in the patient's arm or upper chest will be used for cell infusion. The TIL will be administered over 20-30 minutes at room temperature using a standard infusion protocol or by hanging the infusion bag from a stand and allowing gravity to pull the cells down.

SUMMARY:
The purpose of this protocol is to determine whether autologous TIL infused in conjunction with systemic high-dose IL-2 after non-myeloablative chemotherapy with cyclophosphamide and fludarabine can cause consistent and durable objective responses in patients who have metastatic melanoma at the John Wayne Cancer Institute (JWCI).

ELIGIBILITY:
Inclusion Criteria -

* Patients must have metastatic melanoma with a resectable metastatic lesion of sufficient size and be willing to undergo such a resection for experimental purposes.
* Patients must be > 18 years of age.
* Patients must have measurable disease measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria (in addition to the resected lesion).
* Patients of child bearing potential must agree to use an effective form of birth control during study and up to four months after receiving treatment.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0-1.
* Absolute neutrophil count greater than 1000/mm3 without support of filgrastim.
* Platelet count greater than 100,000/mm3.
* Serum Alanine transaminase/Aspartate transaminase (ALT/AST) less than three times the upper limit of normal.
* Serum creatinine less than or equal to 1.6 mg/dl.
* Total bilirubin less than or equal to 2 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dl.
* Patients must be able to understand and sign the Informed Consent document.

Exclusion Criteria - Tumor/TIL Harvest Exclusion Criteria

* All systemic, cytotoxic therapy (including targeted therapies) must be stopped at least 5 weeks prior to cell infusion (see 2.1.3).
* Women who are pregnant or breastfeeding.
* Life expectancy of less than three months.
* Patients who have received prior treatment with anti-cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibody will be excluded unless a post anti-CTLA-4 antibody treatment colonoscopy was normal with normal colonic biopsies.
* Patients who require immediate active treatment for symptomatic Central Nervous System (CNS) lesions will not be eligible until after treatment of their symptomatic lesions.

Cell Infusion Exclusion Criteria

* Less than 5 weeks has elapsed since any prior systemic therapy at the time the patient receives the preparative regimen. All patients' toxicities must have recovered to a grade 1 or less or as specified in the eligibility criteria in Section 2.1.1. Patients may have undergone minor surgical procedures or focal palliative radiotherapy (to non-target lesions) within the past 5 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria in Section 2.1.1.
* Women of child-bearing potential who are pregnant or breastfeeding.
* Life expectancy of less than three months.
* Systemic steroid therapy more than the equivalent of 10mg/day of prednisone.
* Hemoglobin less than 8g/dl unable to be corrected with transfusion.
* Any active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Any form of primary or secondary immunodeficiency. Must have recovered immune competence after chemotherapy or radiation therapy as evidenced by normal Absolute Neutrophil Count (ANC) > 1000/mm3 and absence of opportunistic infections. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seropositive for HIV antibody.
* Patients with active hepatitis B or active hepatitis C.
* The following patients will be excluded because of inability to receive high dose proleukin:
* Patients will be excluded if they have a history of major EKG abnormalities, symptoms of cardiac ischemia or arrhythmias and have a Left Ventricular Ejection Fraction (LVEF) < 45% on a cardiac stress test (stress thallium, stress Multi Gated Acquisition Scan (MUGA), dobutamine, echocardiogram or other stress test)
* Patients who have a prolonged history of cigarette smoking or symptoms of respiratory dysfunction will be excluded if they have an abnormal pulmonary function test as evidenced by a Forced Expiratory Volume at one second Forced Expiratory Volume at one second (FEV1)< 60% predicted.
* Patients who have received prior treatment with anti-CTLA-4 antibody will be excluded unless a subsequent colonoscopy was normal with normal colonic biopsies (to rule out colitis).
* Patients who require immediate treatment for symptomatic CNS lesions will not be eligible until after treatment of their symptomatic lesions and resolution of symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Faries, MD., FACS, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tumor Infiltrating Lymphocytes (TIL)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: PI left institution prior to completion of enrollment to trial; trial was closed and no analysis of single patient data performed
Arm/Group | Tumor Infiltrating Lymphocytes (TIL)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 21.986 [21.986 to 21.986]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: At the end of 12 week follow up, the proportion of patients that showed clinical response (CR) determined by the disappearance of all target lesions, or partial response (PR) will be calculated. The patient is determined to have partial response as if 30% reduction in the sum of the longest diameter (SLD) of target lesions are shown from the baseline sum LD.
Time Frame: 12 weeks, or until development of new metastases or recurrence
Population: Single patient treated, no formal statistical analysis performed
Measure: Count of Participants; unit: Participants
Arm/Group | Tumor Infiltrating Lymphocytes (TIL)
Number analyzed (Participants) | 1
Participants
  Complete Responder | 0
  Partial Responder | 0
  Non Responder | 1

2. Secondary Outcome: Quality of Life
Description: Quality of Life will be assessed and scored per European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) EORTC-QLQ-C30 version 3.0 requirements. The EORTC QLQ-C30 contains subscales for global health status, and physical, emotional, role, cognitive and social function with higher scores indicating better functioning (19). The change in QOL measured throughout the study period will be examined through mixed effect model adjusting for the baseline. Akaike information criteria (AIC) will be used to determine appropriate covariance structure.
Time Frame: 12 weeks, or until development of new metastases or recurrence
Population: Although the single participant completed a total of 3 surveys, these were never scored or analyzed and data are not available to be reported.
Arm/Group | Tumor Infiltrating Lymphocytes (TIL)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Single patient treated, data collected from baseline up to 72 days.
Arm/Group | Tumor Infiltrating Lymphocytes (TIL)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tumor Infiltrating Lymphocytes (TIL) (N=1)
headache (Nervous system disorders) | 1 (2)
constipation (Gastrointestinal disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (2)
diarrhea (Gastrointestinal disorders) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
facial pain (General disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (2)
White blood cell decreased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
agitation (Psychiatric disorders) | 1 (1) — secondary to PICC line placement and treatment
Other, sunburn (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT02375984/Prot_SAP_000.pdf